CLINICAL TRIAL: NCT00313222
Title: Prospective, Randomized, Placebo-controlled, Double-blind, Multicenter, Parallel Group Study to Assess the Efficacy, Safety and Tolerability of Bosentan in Patients With Inoperable Chronic Thromboembolic Pulmonary Hypertension (CTEPH)
Brief Title: Bosentan Effects in Inoperable Forms of Chronic Thromboembolic Pulmonary Hypertension
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Actelion (Industry)
Responsible Party: Sebastien Roux, MD, Actelion
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: AC-052-366
Record Dates: First submitted 2006-04-10; First posted 2006-04-12 (Estimated); Last update posted 2025-02-03 (Actual); Status verified 2025-01

CONDITIONS: Chronic Thromboembolic Pulmonary Hypertension
Keywords: CTEPH; bosentan
MeSH Terms: interventions — Bosentan

INTERVENTIONS:
Drug: bosentan

SUMMARY:
The present trial investigates a possible use of oral bosentan, which is currently approved for the treatment of symptoms of pulmonary arterial hypertension (PAH), to patients suffering from inoperable chronic thromboembolic pulmonary hypertension (CTEPH) because of (i) peripheral localization of thrombotic material or (ii) persistent or recurrent pulmonary hypertension after pulmonary endarterectomy.

ELIGIBILITY:
Inclusion Criteria:

* Symptomatic pulmonary hypertension in modified NYHA functional class II to IV due to CTEPH as demonstrated by ventilation/perfusion lung scanning and pulmonary angiography.
* CTEPH judged inoperable because of peripheral localization of thrombotic material or persistent or recurrent pulmonary hypertension after pulmonary endarterectomy (PEA) with no evidence of recurrent thromboembolism and not amenable to repeated surgery.
* 6-minute walk test (6MWT) distance < 450 m.
* Hemodynamic evaluation showing: Mean pulmonary arterial pressure (mPAP) >= 25 mmHg; Pulmonary capillary wedge pressure (PCWP) < 15 mmHg; Pulmonary vascular resistance (PVR) at rest >= 300 dyn×sec/cm5
* For patients who underwent PEA, hemodynamic evaluation must have been performed more than 6 months after PEA.
* For all patients, hemodynamic evaluation must have been performed with the 3 months immediately preceding inclusion.
* Men or women >= 18 and =< 80 years of age (Women of childbearing potential must have a negative pre-treatment pregnancy test and use a reliable method of contraception).
* Anticoagulants at efficacious dose for at least 3 months prior to randomization.
* Signed informed consent prior to initiation of any study-mandated procedure.

Exclusion Criteria:

* Other forms of pulmonary hypertension including pulmonary hypertension related to sickle cell disease.
* Obstructive lung disease: FEV1/FVC < 0.5 after bronchodilator.
* Severe restrictive lung disease: Total Lung Capacity < 60% of predicted value.
* Acute or chronic impairment (other than dyspnea), limiting the ability to comply with study requirements (in particular with 6MWT), e.g., angina pectoris, intermittent claudication.
* Symptomatic pulmonary embolism within 6 months prior to randomization.
* Pulmonary endarterectomy within 6 months prior to randomization.
* Psychotic, addictive or other disorder limiting the ability to provide informed consent or to comply with study requirements.
* Illness with a life expectancy of less than 6 months.
* Moderate to severe hepatic impairment, i.e., Child-Pugh Class B or C.
* AST and/or ALT > 3 times the upper limit of normal ranges.· Hemoglobin concentration < 75% the lower limit of normal ranges.
* Pregnancy or breast-feeding.
* Systolic blood pressure (BP) < 85 mmHg.
* Treatment or planned treatment with another investigational drug and/or pulmonary angioplasty within 3 months prior to randomization.
* Treatment with an endothelin receptor antagonist, a phosphodiesterase inhibitor, L-arginine or with prostanoids (excluding acute administration during a catheterization procedure to test vascular reactivity) within 3 months prior to randomization.
* Treatment for pulmonary hypertension within 1 month prior to randomization, excluding calcium channel blockers if present for at least 1 month before randomization.
* Treatment with calcineurin-inhibitors (e.g., cyclosporine A and tacrolimus), sirolimus, fluconazole, glibenclamide (glyburide) within 1 week prior to randomization.
* Known hypersensitivity to bosentan or any of the excipients.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 157 (Actual)
Dates: Start 2005-10; Primary Completion 2007-02 (Actual); Study Completion 2007-03 (Actual)

PRIMARY OUTCOMES:
Change from Baseline to Week 16 in 6-Minute Walk Test distance | Week 16
Change from Baseline to Week 16 in Pulmonary Vascular Resistance at rest | Week 16

SECONDARY OUTCOMES:
Change from Baseline to Week 16 in modified NYHA functional class | Week 16
Time to clinical worsening | Time to clinical worsening

REFERENCES:
- [Derived] Jais X, D'Armini AM, Jansa P, Torbicki A, Delcroix M, Ghofrani HA, Hoeper MM, Lang IM, Mayer E, Pepke-Zaba J, Perchenet L, Morganti A, Simonneau G, Rubin LJ; Bosentan Effects in iNopErable Forms of chronIc Thromboembolic pulmonary hypertension Study Group. Bosentan for treatment of inoperable chronic thromboembolic pulmonary hypertension: BENEFiT (Bosentan Effects in iNopErable Forms of chronIc Thromboembolic pulmonary hypertension), a randomized, placebo-controlled trial. J Am Coll Cardiol. 2008 Dec 16;52(25):2127-34. doi: 10.1016/j.jacc.2008.08.059. PMID 19095129